CLINICAL TRIAL: NCT01768767
Title: Novel Approach of Combined Lithium-Ketamine Therapy in Bipolar Depression: To Preserve Efficacy and Minimize Adverse Effects
Brief Title: Trial of Ketamine and Lithium Therapy in Bipolar Depression
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No funding
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1209010758; T32DA022975 (NIH)
Record Dates: First submitted 2013-01-09; First posted 2013-01-15 (Estimated); Last update posted 2023-03-01 (Actual); Status verified 2020-03

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Ketamine; Lithium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ketamine/Lithium (Experimental): Participant will receive ketamine/lithium
  Interventions: Drug: Ketamine/Lithium
- Ketamine (Active Comparator): Participant will receive ketamine
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Participant will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: Ketamine
  Arms: Ketamine
Drug: Ketamine/Lithium
  Arms: Ketamine/Lithium

SUMMARY:
This study is looking at the safety and efficacy of combined ketamine and lithium therapy for treating patients with bipolar depression who are taking a mood stabilizer that is not working for them.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18-65 years. Females will be included if they are not pregnant and agreed to utilize a medically accepted birth control method (to include oral, injectable, or implant birth control, condom, diaphragm with spermicide, intrauterine device, tubal ligation, abstinence, or partner with vasectomy) or if post-menopausal for at least 1 year, or surgically sterile.
* Able to provide written informed consent according to Yale HIC guidelines.
* Bipolar Disorder in Major Depressive Episode (296.5x or 296.89), as determined by the Structured Clinical Interview for DSM-IV (SCID) patient edition 80
* Montgomery Asberg Depression Rating Scale (MADRS) score of 18 or higher.
* Quick Inventory of Depressive Symptoms - Self-Report (QIDS-SR16) score of 19 or higher.
* Be able to understand and speak English.

Exclusion Criteria:

* Patients with a history of DSM-IV-TR diagnosis of schizophrenia or schizoaffective disorder or currently exhibiting psychotic features associated with their depression.
* Patients with current hypomanic and/or manic symptoms meeting DSM-IV-TR criteria of mixed episode are excluded.
* DSM IV-TR Axis I disorders are excluded if they are considered primary disorders.
* Dementia or suspicion thereof, is also exclusionary.
* Serious suicide or homicide risk, as assessed by evaluating clinician; A serious suicide risk will be considered an inability to control suicide attempts, imminent risk of suicide in the investigator's judgment, or a history of serious suicidal behavior, which is defined using the Columbia-Suicide Severity Rating Scale (C-SSRS) as either (1) one or more actual suicide attempts in the 3 years before study entry with the lethality rated at 3 or higher, or (2) one or more interrupted suicide attempts with a potential lethality judged to result in serious injury or death.
* Substance abuse or dependence during the 3 months prior to screening.
* History of serious medical or neurological illness.
* Signs of major medical or neurological illness on examination or as a result of a 12 lead ECG screening or laboratory studies.
* Abnormality on physical examination. A subject with a clinical abnormality may be included only if the study physician considers the abnormality will not introduce additional risk factors and will not interfere with the study procedure.
* Positive urine drug screen.
* Pregnant or lactating women or a positive urine pregnancy test; for women of childbearing potential.
* Subjects who test positive for HIV or viral hepatitis (hepatitis B and/or C) will be excluded as a means to (1) protect the subjects and research staff from the increased risks of blood borne pathogen transmission during placebo/ketamine infusions and (2) to minimize the factors which might influence the biochemical responses and affect the study outcome. This test will take place at the screening visit. Subjects will be invited back to the Yale Depression Research Program, either for their next study visit or for a HIV/Hep debriefing session. HIV results will be given in a face to face meeting no matter what the results are.
* Patients requiring excluded medications (see Table 3 for details).
* History indicating learning disability or mental retardation.
* Known sensitivity to ketamine or lithium.
* Resting blood pressure lower than 90/60 or higher than 150/90,or resting heart rate lower than 50/min or higher than 100/min.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | 4 Hours to 2 weeks

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptoms - Self-Report (QIDS-SR) | 4 hours to 2 weeks
Clinical Global Impressions Scale (CGI) | 4 hours to 2 weeks

OTHER OUTCOMES:
Young Mania Rating Scale (YMRS) | 4 hours to 2 weeks
Brief Psychotic Rating Scale (BPRS) | 1 and 4 hours
Clinician-Administered Dissociative States Scale (CADSS) | 1 and 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Chadi Abdallah, MD, Principal Investigator — Yale University